CLINICAL TRIAL: NCT04580576
Title: Pilot Study on Gender Differences in Hematopoietic Cell Transplantation Outcomes in the Pediatric Population
Brief Title: Gender Differences in Pediatric Hematopoietic Stem Cell Transplantation (HSCT)
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 25/2019
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: gender, pediatrics, hematopoietic cell transplantation
MeSH Terms: conditions — Coitus | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female group: Pediatric female patients undergoing hematopoietic stem cell transplantation
  Interventions: Procedure: Hematopoietic stem cell transplantation
- Male group: Pediatric male patients undergoing hematopoietic stem cell transplantation
  Interventions: Procedure: Hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Hematopoietic stem cell transplantation — Allogeneic or autologous bone marrow transplant

SUMMARY:
Gender medicine considers the way in which gender, male or female, affects the development and impact of diseases and the response to therapies. It can be said that it is a new transversal dimension of medicine, which evaluates the gender differences in the physiology, pathophysiology and clinic of many diseases and thus sets itself the goal of reaching optimal therapeutic decisions both in men and women based on proven scientific evidence.

Although knowledge of gender medicine has increased significantly in recent years, a gender approach has not been much developed in pediatrics. In the field of bone marrow transplants, hematopoietic stem cell transplantation is known to be the most effective consolidation therapy in some high-risk hematology malignancies such as acute lymphoblastic leukemia and acute myeloid leukemia, and represents one of the potential treatment for patients suffering from solid tumors and genetic hematological, metabolic diseases and primary immunodeficiencies. Huge progress has been made in high resolution donor typing, choice of conditioning regimens, manipulation of hematopoietic stem cells (HSC) and prevention of serious infections in recent years, which have significantly improved the survival rate of patients undergoing to this procedure.

International literature regarding the response and outcomes from hematopoietic cell transplantation in a gender perspective is completely absent, for these reasons this pilot study was born from the need to understand from a broader perspective and in order to better understand how the gender may or not influence the outcome of transplantation in pediatric patients.

This retrospective analysis of the data will concern all patients who underwent allogeneic or autologous bone marrow transplant. The data will be collected from clinical records and from Regional electronic databases. All data will be collected anonymously and an identification code will be assigned to each case.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 4 months and 17 years
2. Diagnosis of oncohaematological disease subjected to hematopoietic stem cell transplantation
3. Allogeneic or autologous bone marrow transplantation from January 2000 to October 2018
4. Consent acquired for the processing of data for research purposes

Ages: 4 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Population of pediatric patients undergoing hematopoietic stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Gender-related difference in overall 12-month toxicity | 12 months after transplant
  Differences in toxicity (hepatic, renal, pulmonary, gastrointestinal) in males and females recipients

SECONDARY OUTCOMES:
Gender difference in overall survival (OS) | 12 months after transplant
  Overall survival comparison from males and females recipients
Gender difference in post-transplant primary disease recurrence | 12 months after transplant
  Incidence of post-transplant leukemic relapse in males and females recipients
Gender difference in the frequency of transplant-related toxicity at 12 months | 12 months after transplant
  Frequency of post-transplant liver, kidney, pulmonary, gastrointestinal, endocrine, cardiac toxicity
Gender difference in infectious complications | 12 months after transplant
  Number of episodes of sepsis / fungal infections / viral reactivations after HSCT
Gender difference in the frequency of adverse events due to pre-transplant conditioning regimen | 12 months after transplant
  Number of chemo- radiotherapy-related adverse events. Toxicity was graded according to National Cancer Institute (NCI) common toxicity criteria
Gender difference in severity of adverse events due to pre-transplant conditioning regimen | 12 months after transplant
  Severity of chemo- radiotherapy-related adverse events. Toxicity wil be graded according to National Cancer Institute (NCI) common toxicity criteria
Gender difference in timing of hematological engraftment | 12 months after transplant
  Engraftment defined as the engraftment of polymorphonuclear neutrophils (PMN) on the first day of 3 consecutive days with PMN number greater than 500 / ml3 and engraftment of platelets defined as number of platelets> 20,000 / ml3 in the absence of platelet transfusion in the previous 5 days.
Gender difference in frequency of primary graft failure | 12 months after transplant
  Engraftment defined as the engraftment of polymorphonuclear neutrophils (PMN) on the first day of 3 consecutive days with PMN number greater than 500 / ml3 and engraftment of platelets defined as number of platelets> 20,000 / ml3 in the absence of platelet transfusion in the previous 5 days.
  Primary graft failure is defined as no evidence of engraftment or hematological recovery of donor cells, within the first month after transplant, without evidence of disease relapse.
Gender difference in frequency of secondary graft failure | 12 months after transplant
  Engraftment defined as the engraftment of polymorphonuclear neutrophils (PMN) on the first day of 3 consecutive days with PMN number greater than 500 / ml3 and engraftment of platelets defined as number of platelets> 20,000 / ml3 in the absence of platelet transfusion in the previous 5 days.
  Secondary graft failure refers to the loss of a previously functioning graft, resulting in cytopenia involving at least two blood cell lineages.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Maestro, PharmD, PhD, Study Director — Institute for Maternal and Child Health IRCCS Burlo Garofolo; Natalia Maximova, MD, Principal Investigator — Institute for Maternal and Child Health IRCCS Burlo Garofolo

IPD SHARING:
Plan to Share IPD: No